CLINICAL TRIAL: NCT01451567
Title: Study That Examined the Effect of a Structured Personalised Ergonomic Intervention Program for Hospital Nurses With Musculoskeletal Complains.
Brief Title: The Effect of a Structured Personalised Ergonomic Intervention for Hospital Nurses With Musculoskeletal Complains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navah Ratzon (Other)
Collaborators: Tel Aviv University (Other); Meir Medical Center (Other)
Responsible Party: Sponsor-Investigator, Navah Ratzon, Head of Occupational Department, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 19505
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2005-05

CONDITIONS: Musculoskeletal Diseases
Keywords: Nurses, Workload, Musculoskeletal System, Intervention
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Musculoskeletal Development

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Ergonomic plan — participants in the intervention group were evaluated by the REBA and received an overall coaching that stretched over four meetings Each session paid special attention to, and included explanations about, the anatomy and physiology of body regions
  Other Names: Ergonomic Intervintion; Musculoskeletal System

SUMMARY:
The purpose of this study is to examine the effect of a structured personalised ergonomic intervention program for hospital nurses with musculoskeletal complains.

DETAILED DESCRIPTION:
In a randomised controlled trial 31 nurses with musculoskeletal complains were observed at work, and an intervention program was completed in 14 nurses with the other 17 acting as controls. The intervention included four meetings during three months. Outcome measures were collected before the intervention and post-tests were gathered three months after the determination of the program.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of half-time work for at least one year
* musculoskeletal pain complaints
* agreement to participate in the interventional study.

Exclusion Criteria:

* Male nurses
* nurses with previously defined job restrictions and
* pregnancy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-06; Primary Completion 2005-10 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Level of stress and control at work, measured by Karasek's questionnaire and Reba | 6 monthes

SECONDARY OUTCOMES:
The prevalence and the level of pain measured by Nordic Questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Netta Abraham Bar-Niv, MA, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel